CLINICAL TRIAL: NCT01092403
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Three-Way Crossover Study to Evaluate the Safety, Tolerability and Clinical Activity of ASM-024 Administered by Inhalation Once Daily to Subjects With Mild Allergic Asthma
Brief Title: Safety, Tolerability and Clinical Activity of ASM-024 in Subjects With Mild Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asmacure Ltée (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ASM-024/II/STA-01
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Mild Allergic Asthma
MeSH Terms: interventions — ASM-024

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASM-024 (Experimental): ASM-024 once daily by inhalation
  Interventions: Drug: ASM-024
- Placebo (Placebo Comparator): Placebo once daily by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASM-024 — ASM-024 50 mg of ASM-024 or 200 mg once daily by inhalation
  Arms: ASM-024
Drug: Placebo — Placebo once daily by inhalation
  Arms: Placebo

SUMMARY:
The study will assess the safety, tolerability and clinical activity of ASM-024 in subjects with mild allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent;
* Male or female subjects, ≥18 years and ≤ 50 years of age;
* Female subjects of childbearing potential must have a negative pregnancy test (serum b-HCG) at Pre-Screening, and a negative urine pregnancy test immediately before the first administration of the study drug for each of the three Treatment Periods. Sexually active females must be willing to use adequate contraception.
* Male subjects must be willing to use a condom with a spermicide for the duration of their participation in the study, plus an additional 30 days following study drug administration and ensure that their partner is using a highly effective method of birth control such as combined oral contraceptives, implants, injectables or a IUD. Male subjects must ensure that their female partner is willing to use adequate contraception;
* Diagnosis of mild allergic asthma that meets the following criteria:

  * Stable on inhaled short-acting beta-2-agonists p.r.n. as the only medication for asthma.
  * Presence of both early asthmatic response (EAR) (at least 20 % fall in FEV1 within 3 hours after allergen inhalation) and late asthmatic response (LAR) (at least 15 % fall in FEV1).
  * Baseline methacholine (PC20) ≤ 16 mg/mL.
* FEV1 of at least 70 % of the predicted value at Pre-Screening and Screening / Baseline;
* BMI ≥ 19 and ≤ 35 kg/m²;
* Body weight ≥ 40 kg;
* Positive skin prick test to at least one common aeroallergen.

Exclusion Criteria:

* Any lung disease other than mild allergic asthma;
* Pregnant or nursing women or women intending to conceive during the course of the study or have a positive serum pregnancy test at Pre-Screening or a positive urine pregnancy test during the study;
* Women of childbearing potential (unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years) not using a highly effective method of birth control. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e., less than 1 % per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence or a partner who has undergone a vasectomy;
* Respiratory tract infections or worsening of asthma within 6 weeks before Screening/Baseline;
* Baseline methacholine PC20 > 16 mg/mL at Screening / Baseline;
* Current cigarette smokers or former smokers with a smoking history of greater than 10 pack years or who stopped smoking within the 12 months preceding enrolment in the study;
* Use of any nicotine containing products within 6 months before Pre-Screening;
* Any of the following concomitant medications:

  * Any medication that are known to prolong QT / QTc interval.
  * Oral or inhaled corticosteroids within 28 days preceding Pre-Screening or systemic corticosteroids within 90 days of Pre-Screening.
  * Long acting beta-2-agonists within one week preceding Baseline.
  * Use of inhaled short-acting β2- agonists or anticholinergics within 8 hours before all study visits to the clinic.
* Known or suspected allergy or sensitivity to nicotine or cholinergic drugs or any drug with similar chemical structure;
* Clinically significant ECG abnormalities at Pre-Screening including clinically significant or marked baseline prolongation of QT / QTc interval (e.g. repeated demonstration of a QTc interval of > 450 ms). Other non clinically significant findings such as sinus bradycardia, sinus arrhythmia, borderline first degree AV block (up to 205 ms), left ventricular hypertrophy (on voltage criteria for a subject less than 40 years old for instance) are permissible if judged to be acceptable by the Qualified investigator;
* Family history of additional risk factors for TdP (e.g., family history of Long QT Syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Late asthmatic response (LAR) | Day 8 of each treatment period
  LAR as measured by the peak drop in FEV1 from 3 to 7 hours post-allergen challenge
Early asthmatic response (EAR) | Day 8 of every treatment period
  EAR as measured by the peak drop in FEV1 from 0 to 3 hours post-allergen challenge
Airway hyperresponsiveness | Days -1, 7 and 9 of each treatment period
  Difference between methacholine PC20 measured 24 hours following allergen challenge and methacholine PC20 measured 24 hours before allergen challenge
Safety and tolerability | Physical examination: Day 9, vital signs: Days -1, 1, 7, 8 and 9; twelve-lead ECG: Days 1, 7, 8 and 9 , AEs throughout the study, safety laboratory assessments Day 1 and 9 and Chest X-Ray: Day 9 of the final treatment period

SECONDARY OUTCOMES:
LAR's FEV1 AUC | Day 8 of every treatment period
  From 3 to 7 hours post-allergen challenge
FEV1 | Day 9
  24 hours post-allergen challenge
EAR's FEV1 AUC | Day 8
  From 0 to 3 hours post-allergen challenge
Change in FEV1 | Days 1, 7, 8 and 9
  Before inhalation of ASM-024 and as soon as possible following inhalation of ASM-024
Induced sputum eosinophil count and eosinophil and neutrophil percentages | Days -1, 7 and 9 of every Treatment Period
Blood eosinophil count | Days -1 and 9 of every Treatment Period
Total and differential WBC count | Days -1 and 9 of every Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (3):
- Canada (3):
  - Mc Master University Health Sciences Center, Hamilton, Quebec
  - Centre de Recherche - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - University of Saskatechewan, Saskatoon, Saskatchewan